CLINICAL TRIAL: NCT06087744
Title: Effects of a Parent-preterm Proximity and Calm Intervention (NeuroN-QI) on the Neurodevelopment of Preterm Infants: A Randomized Pragmatic Clinical Trial
Brief Title: NeuroN-QI: An Intervention to Promote Preterm Infants' Neurodevelopment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Marilyn Aita, Researcher, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MP-21-2023-5375
Record Dates: First submitted 2023-09-13; First posted 2023-10-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Neurodevelopmental Disorders
Keywords: NICU; skin to skin contact; neurodevelopment; preterm infants; positive stimulation; environmental control
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroN-QI (Experimental): Randomized dyads in the experimental group will be asked to do at least one session weekly (ideally 3) skin-to-skin contact (SSC) lasting 2 hours until the age of 36 weeks. Auditory sensory stimulation by mothers or fathers (reading a book) will be carried out during the first 10 minutes during the SSC sessions. The SSC will be followed by a period of calm and rest of one hour during which the infants will rest in their incubator with breast milk's olfactory stimulation. Light and sound control will be done during the entire intervention.
  Interventions: Behavioral: NeuroN-QI
- SSC alone (Active Comparator): Randomized dyads in the control group will be asked to do at least one session weekly (ideally 3) skin-to-skin contact (SPC) lasting 2 hours until the corrected age of 36 weeks. During these sessions, light and noise levels will not be controlled or accompanied of auditory stimulation. SSC periods will not be followed by a calm and rest period with a olfactory stimulation.
  Interventions: Behavioral: SSC alone

INTERVENTIONS:
Behavioral: NeuroN-QI — Skin-to-skin contact (SSC) lasting 2 hours with an auditory sensory stimulation followed by a period of calm and rest of one hour during which the infants will rest in their incubator with breast milk's olfactory stimulation. Light and sound control will be done during the entire intervention.
  Arms: NeuroN-QI
Behavioral: SSC alone — Skin-to-skin contact (SSC) lasting 2 hours
  Arms: SSC alone

SUMMARY:
NeuroN-QI aims to evaluate the effects of an intervention consisting of periods of: 1) parents/preterm infants skin-to-skin contact and auditory stimulation by the parents's voice and 2) calm without manipulation with olfactory stimulation with breast milk in the incubator/bed both combined with appropriate light and noise levels to promote neurodevelopment preterm infants.

ELIGIBILITY:
Inclusion Criteria for preterm infants:

* born between 24 and 33 6/7 weeks GA;
* ready for SSC

Inclusion criteria for mothers and fathers:

* agree to do at least one SSC session/week combined with 10 min of auditory stimulation until 36 weeks of GA of their preterm infant;
* mothers express breast milk for their preterm infants

For twin births (twin pregnancies), fathers will also be invited to participate in the study, so that both infants can participate in the study.

Exclusion criteria for preterm infants:

* congenital anomalies or genetic disorders
* intraventricular hemorrhage > grade II
* are small for GA defined as birth weight <10th percentile
* on postnatal day 19 (maximum days targeted for study start)
* are still receiving analgesics, sedatives, paralyzing agents
* are under mechanical ventilation

Exclusion criteria mothers and fathers:

* are aged <18 years;
* have a physical condition that does not allow the SSC
* abuse illicit substances or alcohol that could influence stress, anxiety and parent- child interactions
* feed their preterm infant exclusively with commercial infant formula
* mothers had a breast surgery that could influence their breast milk production
* do not speak, read or write in French or in English

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopment | 36 weeks gestational age (GA)
  Recording with video and coding with Assessment of Behavioral Systems Organization (ABSO) (from Assessment of Preterm Infant Behavior (APIB))

SECONDARY OUTCOMES:
Neurodevelopment | 4 months and 18 months
  Cerebral discontinuity activity vs. activity with EEG
Neurodevelopment | 4 months and 18 months
  Bayley-IIII (Questionnaire)
Parental Stress | Baseline before randomization and every week after until 36 weeks GA
  Questionnaire - Parental Stress Scale - Neonatal Intensive Care Unit (NICU) (PSS:NICU) - 25 items with a 5-point Likert-type. Minimum value: 25, maximum value: 100. A higher score indicates higher parental stress.
Parental Anxiety | Baseline before randomization and every week after until 36 weeks GA
  Questionnaire - State-Trait Anxiety Inventory (STAI) - 20 items with a 4-point Likert-type scale. Minimum value: 20; maximum value: 80. A higher score indicates higher anxiety.
Parental sensitivity | 4 months ans 18 months
  Recording through videos and coding with Welch Emotional Connection Screen (WECS) - 4 dimensions: mutual attraction, facial communication, vocal communication and sensitivity/reciprocity are coded on a 9-point scale from 1 to 3. Minimum value 4; maximum value 12. Higher scores indicate a better mother-child emotional connection.
Milk production | Every day in mL until study completion at infants' 36 weeks gestational age.
  Through diary
Milk consumption | Total in mL until study completion at infants' 36 weeks gestational age.
  Through charting

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CHU Sainte-Justine, Montreal, Quebec
  - CUSM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No